CLINICAL TRIAL: NCT02692417
Title: Surface Stimulation for Female Sexual Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Bruns (Other)
Responsible Party: Sponsor-Investigator, Timothy Bruns, Assistant Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00101713
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Female Sexual Dysfunction
Keywords: hypoactive desire disorder; female sexual dysfunction; genital arousal disorder; sexual; dysfunction; female; arousal; electrical stimulation; transcutaneous electrical stimulation; women
MeSH Terms: conditions — Coitus | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterior Tibial Nerve Stimulation Group (Experimental): Subjects in this group will have transcutaneous electrical nerve stimulation electrodes placed on the skin surface over their posterior tibial nerve, that is in the area of the ankle, and receive stimulation for 30 minutes in weekly sessions for 12 weeks.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Dorsal Genital Nerve Stimulation Group (Experimental): Subjects in this group will have transcutaneous electrical nerve stimulation electrodes placed on the skin surface over the dorsal genital nerve, that is above and/or on the lateral side of the clitoris, and receive stimulation for 30 minutes in weekly sessions for 12 weeks.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Both arms will receive stimulation from the same TENS (transcutaneous electrical nerve stimulation) unit with identical stimulation frequency, but potentially different amplitudes depending on the subject's stimulation threshold.

SUMMARY:
Female sexual dysfunction, including sexual arousal disorder, has a significant clinical impact, affecting millions of women in the United States alone. Peripheral nerve stimulation, such as posterior tibial nerve stimulation (PTNS) and dorsal genital nerve stimulation (DGNS) can modulate neural circuits for bladder and fecal continence. The investigators hypothesize that periodic DGNS and PTNS will modulate autonomic neural circuits and promote improvements in sexual function in women with sexual arousal disorder. Subjects will be randomized to receive one of the stimulation approaches. Subjects will have weekly 30-minute sessions across twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥ 18 years of age
* Sexually active ≥ 1 time per month (≥ 2 times per month preferred)
* Score of 19 or less on a 6-question set of the Female Sexual Function Index (FSFI) survey
* Neurologically stable
* Ambulatory
* Capable of giving informed consent
* English speaking
* Capable and willing to follow study procedures

Exclusion Criteria:

* Men
* Women ≤ 17 years of age
* Pregnant or planning to get pregnant during the study period
* Clinically diagnosed neurological bladder dysfunction
* Prior experience with PTNS or DGNS
* Current use of transcutaneous electrical nerve stimulation (TENS) on pelvis, back, or legs
* Implanted pacemaker, defibrillator, spinal cord stimulator, or sacral root stimulator
* Taking flibanserin
* Taking any investigational drug
* History of neurologic diseases or impairments
* Any other factors that the investigators feel would place the patient at increased risk from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bruns, PhD, Principal Investigator — University of Michigan; Mitchell Berger, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posterior Tibial Nerve Stimulation Group | Dorsal Genital Nerve Stimulation Group
Started | 9 | 7
Completed | 3 | 6
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject enrolled in the PTNS arm did not complete the initial survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Posterior Tibial Nerve Stimulation Group | Dorsal Genital Nerve Stimulation Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (14.3) | 46.6 (14.8) | 40.9 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 6 | 10
  Black | 1 | 0 | 1
  Asian or Pacific Islander | 0 | 1 | 1
  Other | 3 | 0 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.5) | 26.5 (4.5) | 26.8 (4.4)
Relationship Status [Count of Participants; unit: Participants]
  Single | 1 | 1 | 2
  Nonmarried relationship | 2 | 1 | 3
  Married | 5 | 5 | 10
On prescription antidepressant [Count of Participants; unit: Participants] | 3 | 3 | 6
Baseline FSFI [Mean (Standard Deviation); unit: score on a scale] — The Female Sexual Function Index (FSFI) is a validated, 19-item questionnaire evaluating sexual functioning in women. A clinical cutoff score of 26.55 differentiates women with and without sexual dysfunction, with below a 26.55 indicating sexual dysfunction. The minimum score one can receive is 2, and the maximum score is 36. Higher scores indicate better sexual functioning. The total FSFI score is the sum of the six subcategories (desire, arousal, lubrication, orgasm, satisfaction and pain) which each have a maximum score of 6.
  score on a scale | 18.4 (5.1) | 16.0 (5.3) | 17.3 (5.2)
Baseline SF-36 [Mean (Standard Deviation); unit: units on a scale] — The 36-Item Short Form Health Survey (SF-36) evaluates quality of life. The minimum score is 0 and the maximum score is 100, with lower scores representing lower quality of life.
  units on a scale | 78.8 (15.3) | 87.4 (4.2) | 82.8 (12.0)
Baseline AUASI [Mean (Standard Deviation); unit: units on a scale] — The 7-question American Urological Association Symptom Index (AUASI) bladder symptom index evaluates bladder functioning. Lower scores indicate better urological function. There is a minimum score of 1 and a maximum score of 35.
  units on a scale | 8.6 (6.4) | 4.6 (2.6) | 6.7 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: 6 Weeks - Total FSFI Score
Description: Sexual function was measured by the Female Sexual Function Index (FSFI), which is a validated, 19-item questionnaire evaluating sexual functioning in women. A clinical cutoff score of 26.55 differentiates women with and without sexual dysfunction, with below a 26.55 indicating sexual dysfunction. The minimum score one can receive is 2, and the maximum score is 36. Higher scores indicate better sexual functioning. The total FSFI score is the sum of the six subcategories (desire, arousal, lubrication, orgasm, satisfaction and pain) which each have a maximum score of 6. Each subcategory has questions scored either 0-5 (arousal, lubrication, orgasm, pain) or 1-5 (desire, satisfaction). The sum for each subcategory is multiplied by a factor of either 0.3 (arousal, lubrication), 0.4 (orgasm, satisfaction, pain) or 0.6 (desire). The minimum score for desire is 1.2 and for satisfaction is 0.8, the rest are 0. Only the results from the 9 subjects who completed the study were analyzed.
Time Frame: 6 weeks after beginning of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Tibial Nerve Stimulation Group | Dorsal Genital Nerve Stimulation Group
Number analyzed (Participants) | 3 | 6
score on a scale | 26.0 (7.8) | 17.4 (6.6)
Statistical Analysis 1: Comparison: Posterior Tibial Nerve Stimulation Group; Wilcoxon signed rank test comparing FSFI score from baseline to time point; Test type: Other; p = 0.109, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dorsal Genital Nerve Stimulation Group; Wilcoxon signed rank test comparing FSFI score from baseline to time point; Test type: Other; p = 0.225, Wilcoxon (Mann-Whitney)

2. Primary Outcome: 12 Weeks - Total FSFI Score
Description: as for outcome 1
Time Frame: 12 weeks after beginning of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Tibial Nerve Stimulation Group | Dorsal Genital Nerve Stimulation Group
Number analyzed (Participants) | 3 | 6
score on a scale | 27.8 (4.8) | 18.7 (6.9)
Statistical Analysis 1: Comparison: Posterior Tibial Nerve Stimulation Group; Wilcoxon signed rank test comparing FSFI score from baseline to time point; Test type: Other; p = 0.109, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dorsal Genital Nerve Stimulation Group; Wilcoxon signed rank test comparing FSFI score from baseline to time point; Test type: Other; p = 0.046, Wilcoxon (Mann-Whitney)

3. Primary Outcome: 18 Weeks - Total FSFI Score
Description: as for outcome 1
Time Frame: 18 weeks after start of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Tibial Nerve Stimulation Group | Dorsal Genital Nerve Stimulation Group
Number analyzed (Participants) | 3 | 6
score on a scale | 26.2 (8.6) | 18.8 (5.4)
Statistical Analysis 1: Comparison: Posterior Tibial Nerve Stimulation Group; Wilcoxon signed rank test comparing FSFI score from baseline to time point; Test type: Other; p = 0.109, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dorsal Genital Nerve Stimulation Group; Test type: Other; p = 0.028, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected until the final survey (18 weeks after start of stimulation) was collected.
Arm/Group | Posterior Tibial Nerve Stimulation Group | Dorsal Genital Nerve Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/9 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posterior Tibial Nerve Stimulation Group (N=9) | Dorsal Genital Nerve Stimulation Group (N=7)
Sciatic Nerve Pain (Nervous system disorders) | 1 (1) | 0 (0) — Subject had a history of sciatic pain and aggravation reemerged during stimulation

LIMITATIONS AND CAVEATS:
There were challenges in recruitment and retention for the study. Six of the seven subjects who discontinued the study were in the PTNS arm, leading to an unequal distribution of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT02692417/Prot_SAP_000.pdf